CLINICAL TRIAL: NCT06350409
Title: Adolescent Outcomes of Post-operative Opioid EXposure
Acronym: APEX
Status: Recruiting | Type: Observational
Sponsor: Sharon Levy (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Levy, Chief, Division of Addiction Medicine, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Other Study IDs: CTN-0146; UG1DA015831-22S4 (NIH); 3UG1DA015831-24S1 (NIH)
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder; Pain, Chronic
Keywords: Adolescent Opioid Use; Post operative pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to examine the factors associated with the transition from medical exposure to opioids with "signposts" of future opioid use disorder among adolescent surgical patients. The main question aims to identify factors (moderators, mediators, and covariates) associated with risk factors for opioid use disorder (ROUD) in the 12 months following major surgery with opioid exposure among adolescents aged 12-17. Participants will be asked to complete electronic surveys pre- and post-operatively and approve the collection of peri-operative data from the Electronic Medical Record to assess correlations.

DETAILED DESCRIPTION:
This project will collect data from a diverse sample of 10,000 dyads, including adolescent (aged 12-17 years, inclusive) patients undergoing major surgery with planned post-operative opioid analgesic use. and a parent (Total N=20,000) to identify ROUD that may occur within the 12 months after surgery. The resulting data repository will allow clinician scientists and physicians to develop research-informed pain management protocols for adolescent surgical patients to reduce the risk of OUD in this vulnerable population.

Using a novel combination of data sources (electronic medical records (EMR), patient-reported outcomes, and parent-reported outcomes), this study investigates the twin problems of postoperative pain and ROUD in adolescent surgical patients. Using real-world evidence to evaluate longitudinal behaviors and outcomes.

This project will provide insights into the associations between post-operative pain management and ROUD in adolescents. Findings could yield information about potential risks, which may inform future studies and ultimately lead to new screening tools to assess risk before opioid prescribing, updated protocols for managing pain intra-operatively and post-operatively in high-risk populations, updated patient and family education materials to reduce risks for those undergoing painful procedures, and revised recommendations for monitoring for patients being treated for pain. Furthermore, the project enables the establishment of an infrastructure among pediatric surgical centers that can be used for future projects to evaluate the best postoperative outcomes for youth.

Aim 1: Determine the frequency of ROUD. Because this is a novel measure of ROUD, we will use the first 1,000 samples to estimate the incidence of ROUD developing among adolescents in the year following surgery with post-operative opioid analgesia.

Aim 2: We will use machine learning models to develop and validate screening algorithms designed to detect "early warning signs" or Risk factors for Opioid Use Disorder (ROUD). The features in these models will include the pre-, intra- and postoperative EMR-derived data elements, as well as the survey data. We will fit the models against the primary outcome described above. Model evaluation will be done via cross-validation, where the models will be fit on a randomly selected training set of patients and evaluated on the remaining held-out subset of the patients to be used exclusively for testing the performance of the final models.

Aim 3: Developing and validating a prediction model designed to predict a clinical trajectory of post-surgical opioid use and pain. We will use clustering to identify typical patient trajectories of opioid use, and we will use similar prediction and validation techniques as in Aim 1 to build a prediction model for these trajectories.

ELIGIBILITY:
Adolescent Inclusion Criteria

1. Adolescents between the ages of 12 to 17 years old, inclusive, who are scheduled to undergo a scheduled surgical procedure with a greater than 90% likelihood of requiring opioid analgesia for at least 48 hours post-operatively (as an inpatient) or discharged home with at least a 48-hour supply of prescription opioids.

   • Opioid prescribing practices vary by institution; therefore, eligible surgical procedures will be determined on a site-by-site basis.
2. Adolescents willing and able to provide informed assent and have a parent/caregiver willing to provide informed consent.

Parent/Caregiver Inclusion Criteria

1. Parent or legal guardian of an eligible adolescent.
2. Parent or legal guardian willing and able to provide written informed consent.

Adolescent Exclusion Criteria

Adolescents meeting any of the following criteria will be excluded from study participation:

1. Adolescents who have been prescribed opioids in the past 2 years for pain due to a chronic medical condition.
2. Adolescents who have a current chronic medical condition that requires ongoing opioid pain management and treatment such as sickle cell disease, arthritis, or cancer.
3. Adolescents who do not have a caregiver who is willing to co-participate in the study.
4. Adolescents who cannot speak or read English at a 4th-grade level as determined by medical or research staff.
5. Adolescents who are currently in the custody of the Department of Youth Services, jail/prison, or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities.
6. Adolescents who are currently in the custody of the Department of Children and Families or living with a foster family.
7. Adolescents who are currently pregnant or parenting.
8. Adolescents that self or parent report of ever having been diagnosed with opioid use disorder, or prescribed buprenorphine, methadone, or naltrexone to treat opioid use disorder.
9. Adolescents who are currently enrolled in an intervention study that aims to impact opioid prescription or pain management pre-, peri-, or post-operatively.

Parent/Caregiver Exclusion Criteria

Parents/Caregivers meeting any of the following criteria will be excluded from study participation:

1. Parents/Caregivers who cannot speak or read English or Spanish at a 4th grade level as determined by medical or research staff.
2. Parents/Caregivers that are currently incarcerated.
3. Parents/Caregivers that are in physical or mental distress that precludes study participation as determined by clinical or study staff.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study aims to recruit a convenience sample of approximately 10,000 dyads of adolescent (12-17 years, inclusive) patients and one parent (Total N=20,000). Adolescent participants will be undergoing scheduled surgeries with a greater than 90% likelihood of requiring opioid analgesia for at least 48 hours post-operatively (as an inpatient) or discharged home with at least a 48-hour supply of prescription opioids.
  Opioid prescribing practices vary by institution; therefore, eligible surgical procedures will be determined on a site-by-site basis. Exemplar surgeries at BCH and CCHMC sites include spinal fusion surgery, Nuss procedure, and anterior cruciate ligament reconstruction. Both inpatient and outpatient surgical procedures will be considered.
  All adolescent participants will be aged 12-17 at the time of enrollment and are children as defined by the NIH Policy on I
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Risk of opioid use disorder due to prolonged pain that develops within the first year after surgery. | 12 months
  The patient self-report an average pain score of more than 3/10 in the last 7 days on the Brief Pain Inventory (BPI) at 3 or more months postoperatively.
Risk of opioid use disorder due to prolonged opioid use that develops within the first year after surgery. | 12 months
  Any adolescent self-report or parent report of opioid medication use more than 3 or more months postoperatively.
Risk of opioid use disorder due to postoperative non-medical use of prescription opioids (NMUPO) that develops within the first year after surgery. | 12 monhts
  Any adolescent self-report or parent report of use of opioid medication that is > than prescribed, or more frequently than prescribed, or not prescribed to the adolescent.
Risk of opioid use disorder due to increased rate of change in substance use that develops within the first year after surgery. | 12 month
  Adolescent self-report of rate of increase of substance use frequency greater than the 75th percentile of an age- and sex-matched cohort compared to nationally representative data
Risk of opioid use disorder due to post-surgical trauma that develops within the first year after surgery. | 12 months
  Adolescent self-report of post-surgical trauma and stress as measured by >11 on the Child PTSD Symptom Scale (CPSS) 3 or more months postoperatively.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Boston Childrens Hopsital - Division of Addiction Medicine, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: APEX study information website — https://www.childrenshospital.org/research/labs/adolescent-outcomes-post-operative-opioid-exposure-research